CLINICAL TRIAL: NCT05577611
Title: An Open, Single Center, Randomized Controlled Clinical Study of UCB (Cord Blood) in the Treatment of Newly Diagnosed Acute Myeloid Leukemia (AML)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Principal Investigator, Fuling Zhou, Chief physician, Zhongnan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCBT
Record Dates: First submitted 2022-09-09; First posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: UCB (Cord Blood) Microtransplantation in the Treatment of Newly Diagnosed Acute Myeloid Leukemia (AML)
Keywords: acute myeloid leukemia; cord blood; HSCT
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Basic chemotherapy + UCB transplantation (Experimental)
  Interventions: Combination Product: Basic chemotherapy + UCB transplantation

INTERVENTIONS:
Combination Product: Basic chemotherapy + UCB transplantation — The basic chemotherapy regimen was the same as that of the control group
  UCB micro transplantation scheme:
  Aza 100mg, 75mg/m2/d, IVGTT, D-10 to D-4
  Ara-C 1000mg/m2/q12h, IVGTT, D-3 to D-2
  Single non consanguineous umbilical cord blood (NC > 1.5 * 10 ^ 7 / kg), IVGTT, D0
  Bone marrow aspiration smear, MRD and bone marrow chimerism were detected on D14, d30 and D60 after transplantation.

SUMMARY:
In recent years, the curative effect of AML has been greatly improved. However, 20% - 30% of young patients and 40% - 50% of old patients will relapse again. Its re induction response rate is low, the survival period is short, and the prognosis is very poor. At present, there is no standard treatment scheme. Although a small number of patients can benefit from allogeneic hematopoietic stem cell transplantation (allo HSCT), most patients lack suitable donors. The choice of high-dose chemotherapy is a rescue treatment scheme, but the treatment-related hematology or non hematology related toxicity and high mortality make the scheme controversial, especially for the elderly. Some studies have proposed a new treatment method combining chemotherapy with peripheral blood hematopoietic stem cell infusion after mobilization of HLA mismatched donors. Preliminary clinical studies verified that after more than 70 cases of elderly acute myeloid leukemia were treated with microtransplantation, the complete remission rate reached 80%, the 2-year disease-free survival rate reached 39%, the early mortality rate was only 6.7%, and the median recovery time of neutrophils and platelets was 11 and 14.5 days, respectively, which was significantly different from the control group of chemotherapy alone. After that, the micro transplantation technology was extended to the treatment of myelodysplastic syndrome and lymphoma, and good results were also obtained. Compared with peripheral blood / bone marrow hematopoietic stem cells, umbilical cord blood (UCB) hematopoietic stem cells have the advantages of rapid access, convenient source, no harm to donors, and low requirements for HLA matching. The immune cells in cord blood hematopoietic stem cells are mostly Na ï ve and immature immune cells, so the incidence and severity of graft-versus-host disease (GVHD) after unrelated cord blood transplantation are low, which not only reduces the failure of transplantation due to GVHD, but also avoids a series of complications and high costs brought by complex GVHD prevention and treatment techniques. Because cord blood is rich in CD16 + CD56 + NK cells and CD3 + T cells, cord blood hematopoietic stem cell transplantation also plays an important role in GVL.

ELIGIBILITY:
Inclusion Criteria:

* No previous transplantation treatment;
* Acute myeloid leukemia;
* Karnofsky score ≥ 60%, physical strength status of Eastern Cooperative Oncology Group (ECoG) ≤ 2;
* Cord blood with HLA matching 0-3 / 6 and blood type matching;

Exclusion Criteria:

* Second-class or above surgery within 4 weeks before randomization;
* Currently diagnosed as malignant tumor other than AML or under treatment;
* Acute promyelocytic leukemia, myeloid sarcoma, chronic myeloid leukemia accelerated phase and acute transformation phase;
* Stroke or intracranial hemorrhage occurred within 6 months before randomization;
* Uncontrolled or symptomatic arrhythmias;
* Congestive heart failure;Myocardial infarction within 6 months before screening;
* Any grade 3 (moderate) or grade 4 (severe) heart disease (according to NYHA);
* Active human immunodeficiency virus (HIV) or active hepatitis B virus (HBV) Dependence on illicit drugs;
* Mental or cognitive impairment;
* Participate in other clinical trials 1 month before registration;

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2022-08-10 (Actual); Primary Completion 2024-12-25 (Estimated); Study Completion 2024-12-25 (Estimated)

PRIMARY OUTCOMES:
Change from marrow blast in percentage at Week 18 | Day 0，Day 1，Week 1，Week4，Week 12，Week 18
  marrow blast in percentage
Change from Blood routine in plasma at Week 18 | Day 0，Day 1，Week 1，Week4，Week 12，Week 18
  WBC
Change from Blood routine in plasma at Week 18 | Day 0，Day 1，Week 1，Week4，Week 12，Week 18
  RBC
Change from Blood routine in plasma at Week 18 | Day 0，Day 1，Week 1，Week4，Week 12，Week 18
  PLT
Change from liver and kidney function at Week 18 | Day 0，Day 1，Week 1，Week4，Week 12，Week 18
  ALB
Change from liver and kidney function at Week 18 | Day 0，Day 1，Week 1，Week4，Week 12，Week 18
  GLB
Change from liver and kidney function at Week 18 | Day 0，Day 1，Week 1，Week4，Week 12，Week 18
  eGFR
ECG QT Interval，ST segment，P wave，QPS wave group | Day 1
  We will record this index in the first day
Change from Blood routine in plasma at Week 18 | Day 0，Day 1，Week 1，Week4，Week 12，Week 18
  Hb
Change from liver and kidney function at Week 18 | Day 0，Day 1，Week 1，Week4，Week 12，Week 18
  Creatine
Change from liver and kidney function at Week 18 | Day 0，Day 1，Week 1，Week4，Week 12，Week 18
  β2-MG

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided